CLINICAL TRIAL: NCT02696408
Title: Efficacy of Prophylactic Low Level Laser Therapy (LLLT) Performed by Nurses for Decreasing Severity of Oral Mucositis During Hematopoietic Stem Cell (HSC) Transplantation : a Randomized Double Blind Multicenter Prospective Phase III Trial
Brief Title: Efficacy of Prophylactic Low Level Laser Therapy (LLLT) Performed by Nurses for Decreasing Severity of Oral Mucositis During Hematopoietic Stem Cell (HSC) Transplantation
Acronym: STOP MUCITES
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Institut de Cancérologie de la Loire (Other)
Collaborators: Hospices Civils de Lyon (Other); Centre Leon Berard (Other); Société Biophoton (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2015-07; 2015-A01492-47 (Other: ANSM)
Record Dates: First submitted 2016-02-25; First posted 2016-03-02 (Estimated); Last update posted 2020-01-29 (Actual); Status verified 2020-01

CONDITIONS: Hematologic Malignancy
Keywords: Mucositis; Low level laser therapy; Autograft; Allograft
MeSH Terms: conditions — Hematologic Neoplasms; Mucositis | interventions — Laser Therapy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Laser treatment (Experimental): preventive treatment performed by nurses of mucositis by laser treating daily by scanning the entire oral cavity for 2 minutes with a power of 250 mW associated with mouthwashes several times a day (standard preventive treatment of mucositis)
  Interventions: Device: Laser treatment
- laser-off (Placebo Comparator): daily laser-off session performed by nurses associated with mouthwashes several times a day (standard preventive treatment of mucositis)
  Interventions: Device: Placebo

INTERVENTIONS:
Device: Laser treatment — Patients randomized to the experimental arm receive in addition to mouthwash, preventive treatment of mucositis by LLLT performed by nurses consisting of daily scanning the entire oral cavity for 2 minutes with a power of 250 mW, starting with conditioning and ongoing until the onset of mucositis of grade 1.
  If the mucositis is localised, preventive laser will be kept on the healthy zones, and curative laser will be performed on painful zone. If the mucositis is general (more than 1 site), preventive laser is stopped for curative laser only.
  Other Names: Oncolase DIGI D5W200
  Arms: Laser treatment
Device: Placebo — Patients randomized to the Placebo arm receive in addition to mouthwash fictive laser treatment performed by nurses until the onset of mucositis of grade 1.
  If the mucositis is localised, fictive laser will be kept on the healthy zones, and curative laser will be performed on painful zone. If the mucositis is general (more than 1 site), fictive laser is stopped for curative laser only.
  Arms: laser-off

SUMMARY:
The LLLT has an anti-inflammatory, analgesic effect and accelerates the healing of ulcerated lesions. There are little data in the literature showing its efficacy in prevention of mucositis in cohorts of patients with hematopoietic stem cells transplantation.

The main objective of this study is to assess the efficacy of a prophylactic low level laser therapy performed by nurses on the severity of oral mucositis during HSCT.

DETAILED DESCRIPTION:
The main end point for efficacy is the reduction of severe mucositis (grade 3 or more). The secondary efficacy endpoints are the reduction of mucositis, whatever the grade, the reduction of time with mucositis, the time to onset of mucositis symptoms, the reduction of pain intensity and evaluation of quality of life.The secondary endpoints for safety are severe adverse events and potential toxicity. Patients will be allocated at inclusion with a 1/1 ratio either to laser-on or laser-off groups. In the laser group, patients will undergo laser therapy performed by nurses, which will consist of irradiation of the whole oral cavity during 2 minutes with 250mW power. In the laser-off group, laser therapy will be carried out with equipment off during the same time, and still performed by nurses. Protective eye shields will be used to avoid detrimental effects on eyes and to keep the subjects blind.

ELIGIBILITY:
Inclusion Criteria:

* Patient undergoing autologous or allogeneic HSC (Hematopoietic Stem Cell) transplantation with myeloablative conditioning
* Patient affiliated to a social security
* Signed inform consent

Exclusion Criteria:

* Patient undergoing HSCT (Hematopoietic Stem Cell Transplantation) with reduced intensity conditioning Slavin (FB2) or Seattle (F-2 Gy TBI)
* Protected major patient
* Pregnant woman
* Patient with pacemaker
* Epileptic Patient

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 234 (Actual)
Dates: Start 2016-06-27 (Actual); Primary Completion 2019-11-07 (Actual); Study Completion 2019-12-09 (Actual)

PRIMARY OUTCOMES:
prevalence of grade 3 mucositis and more | 30 days
  prevalence of grade 3 and more mucositis following the classification proposed by WHO (world health organization)

SECONDARY OUTCOMES:
number of all grades of mucositis | 30 days
  The number of all grades of mucositis will be reported at day 30 post graft for all patients.
duration of mucositis | 30 days
  The duration of mucositis will be reported at day 30 post graft for all patients.
time of onset of mucositis | 30 days
  time of onset of mucositis will be assessed by measuring the interval between the beginning of packaging and the first day of mucositis has been assessed at a grade 1
Pain | 30 days
  Pain will be reported for each patient during their participation: 30 days post graft maximum.
Quality of life | 30 days
  Quality of life will be reported for each patient during their participation: 30 days post graft maximum.
Safety | 30 days
  serious adverse events will be reported for each patient during their participation: 30 days post graft maximum.

CONTACTS AND LOCATIONS:
Overall Officials: Emmanuelle TAVERNIER, MD, Principal Investigator — Institut de Cancérologie Lucien Neuwirth
Locations (3):
- France (3):
  - Centre Léon Bérard, Lyon
  - Centre Hospitalier Lyon Sud, Pierre-Bénite
  - Institut de Cancérologie Lucien Neuwirth, Saint-Priest-en-Jarez

IPD SHARING:
Plan to Share IPD: No